CLINICAL TRIAL: NCT02358434
Title: Kinematics Analysis: Cruciate Retaining, Fixed Bearing Primary Total Knee Arthroplasty With the ATTUNE TM Knee System
Brief Title: ATTUNE TM Video-fluoroscopy Study
Status: Completed | Type: Observational
Sponsor: Dr. Renate List (Other)
Responsible Party: Sponsor-Investigator, Dr. Renate List, Dr. sc. ETH Zurich, Institute for Biomechanics, ETH Zürich
Organization: Institute for Biomechanics, ETH Zürich (Other)
Other Study IDs: ATTUNE-2015
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Total Knee Arthroplasty
Keywords: Implant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Observational use of fluoroscopy

SUMMARY:
The proposed study is a retrospective, observational study. A group of 5 subjects with the AttuneTM cruciate retaining (CR) fixed bearing total knee arthroplasty (TKA) are analysed during level walking, a deep knee bend, sitting down onto a chair, standing up from a chair and stair descent at least 12 months post-operatively, in terms of 3D fluoroscopic assessed tibio-femoral TKA motion as well as simultaneous skin marker assessed whole leg motion and ground reaction forces. The obtained information helps the manufacturer (DePuy) to evaluate, bring to market and advance the implant. Furthermore the information will be integrated in a model, which will be developed at the Center for Orthopaedic Engineering, University of Denver. By means of this model, different conditions such as the use of an advanced prosthesis design can be simulated and tested.

The objective of this study is in a first step to demonstrate the capability of data collection and analysis of level gait, deep knee bend, sitting down onto a chair, standing up from a chair and stair descent on a limited sample size of five subjects. Secondly to quantify and describe the three-dimensional kinematics for the cruciate retaining (CR), fixed bearing AttuneTM TKA during daily activities such as those mentioned.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral TKA (ATTUNETM) due to osteoarthrosis (OA)
* Body mass index (BMI) ≤ 33
* Good clinical outcome, Knee injury and Osteoarthritis Outcome Score (KOOS) > 70
* No or very low Visual Analog Scale for Pain (VAS) < 2
* At least one year post-op
* Standardized general health survey score (SF-12) within the normal range for people in their age group

Exclusion Criteria:

* Actual significant problem on lower extremities
* Misaligned TKA
* Any other arthroplasty at the lower extremities
* Patient incapable to understand and sign informed consent
* Incapable of performing the motion tasks
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prof. Dr. med. Carsten Perka will do the recruitment, since he is the surgeon that worked the most with this implant and therefore also has the biggest population of possibly eligible patients. Furthermore the patients already know and trust him, which could lead to a greater success in the recruitment as well. For these reasons the financial source DePuy Synthes, Johnson and Johnson, requires that the clinical collaborator Prof. Dr. med. Carsten Perka will do the recruitment. He works in the Charité in Berlin, Germany, where he does the recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Relationship between the knee flexion angle and the medial and lateral anterior-posterior translation of the condyles | 3 hours
  The primary outcome of this pilot study is the relationship between the knee flexion angle and the medial and lateral anterior-posterior translation of the condyles during level walking, stair descent, standing up from a chair, sitting onto a chair and deep knee bend.

CONTACTS AND LOCATIONS:
Overall Officials: Renate List, PhD, Principal Investigator — ETH Zurich
Locations (1):
- Institute for Biomechanics, Zurich, Canton of Zurich, Switzerland